CLINICAL TRIAL: NCT04524377
Title: Evaluation of the Influence of Deep Brain Stimulation on the Spinal Deformities Associated With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Spindler, Dr. med. Philipp Spindler, Resident, Principal Investigator, Charite University medicine / department of neurosurgery, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40000256
Record Dates: First submitted 2020-08-14; First posted 2020-08-24 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease; Spine Degeneration; Spine Deformity; Spinal Disease
Keywords: Deep Brain Stimulation; Parkinson Disease; Spine
MeSH Terms: conditions — Parkinson Disease; Spinal Diseases | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Deep Brain Stimulation (DBS) of the Nucelus subthalamicus (STN) in patients with Parkinson's Disease (PD).
Masking Description: The Radiologist who evaluated X-rays ist masked regarding timepoint of investigation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS for Parkinsons Disease (Experimental)
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Deep brain stimulation involves implanting electrodes within certain areas of the brain. These electrodes produce electrical impulses that regulate abnormal impulses. Or the electrical impulses can affect certain cells and chemicals within the brain.
  The amount of stimulation in deep brain stimulation is controlled by a pacemaker-like device placed under the skin in the upper chest. A wire that travels under the skin connects this device to the electrodes in the brain.

SUMMARY:
The intention of the study is to investigate whether Deep Brain Stimulation (DBS) will improve postural deformities of patients with Parkinson's disease.

DETAILED DESCRIPTION:
1. Introduction

   Postural deformities are frequent comorbidities that limit the quality of life in patients with Parkinson's disease. Subject of the study is the investigation of postural deformities as a concomitant disease in connection with therapy with DBS. The aim of this prospective study is to examine the effect of deep brain stimulation on postural instability and thus the quality of life of patients.
2. Study outline

   The aim of this prospective study is to investigate the effect of DBS on postural instability and thus the quality of life of patients.

   For this purpose, the investigators would like to evaluate 50 participants before and at certain time points (three, six, twelve and 24 months) after DBS surgery. X-rays of the entire spine are carried out using EOS® technology and biodynamic measurements of the spine using the Epionics SPINE ® system. In addition, the Investigators collect the 39-item PD Questionnaires (PDQ-39), Unified Parkinson's Disease Rating Scale (UPDRS) Part III, Visual Analog Scale (VAS) and Oswestry Disability Index (ODI) as clinical parameters.

   Our hypotheses (I): DBS improves the sagittal balance of the spine and the pelvic rotation as a corresponding compensation mechanism for this incorrect posture (II) The participant's mobility improves in course of DBS in terms of scope and speed (III) In course after DBS, back pain is significantly reduced and the participant's everyday life is easier to cope with.

   The investigators hope to gain new insights into the pathophysiology of the spinal deformities associated with Parkinson's disease from the study and to expand the indication for DBS to include clinically relevant spinal complaints.
3. Consent to the study

   The study was positively assessed by the Charité ethics committee and the Federal Office for Radiation Protection.

   Consent for study inclusion is sought after explanation and agreement to DBS treatment for participants with Parkinson's disease. Thus, participants capable of consenting to the DBS treatment get the study details explained themselves and may or may not agree to participate. If a participant is incapable for consenting to the proposed treatment, he may not be enrolled in the study.
4. Safety of DBS for Parkinson's disease and further risks for participants

   Deep brain stimulation is a well-established and well-tolerated treatment for Parkinson's disease.

   The study-related risks result from the multiple X-ray examinations of the spine (effective dose 2.6 µSv per examination). There are no other study-related risks of the planned ones.
5. Insurance Coverage

An insurance was taken out for all study participants who took part in this study at HDI-Gerling Industrie Versichung AG, Riethorst 2, 30659 Hanover, Insurance number: 5701032603017.

German laws §§ 40 to 42 Arzneimittelgesetz or §§ 20 to 23 Medizinproduktegesetz are not applicable.

The Investigators are insured against fault-based damage through the existing liability insurance of their clinic.

ELIGIBILITY:
Inclusion Criteria:

* women and men, over 18 years of age
* medical indication for deep brain Stimulation for Parkinson's Disease
* signed declaration of consent

Exclusion Criteria:

* withdrawal of consent
* non-Parkinson's-associated diseases of the spine
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Sagittal Imbalance | Two years after DBS
  Sagittal vertical axis (SVA) in X-Ray of the Spine. SVA is identified as the location of the head with respect to the normal center of gravity by a plumb line dropped from the center of the C7 vertebral body to the posterior superior corner of the sacral end plate. It is measured in cm with pathological values >5cm and sagital Imbalance defined as SVA >10cm.

SECONDARY OUTCOMES:
Spine Mobility | Two years after DBS
  Function of the back as well as the position and movement of the pelvis in patients with Parkinson's disease with a non-invasive measuring system, (Epionics SPINE System®). Scope (in degrees) and speed (in degrees/s) of motion are measured.
Oswestry Disability Index (ODI) | Two years after DBS
  The Oswestry Disability Index (ODI) questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered summed up and multiplied by two. To obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Visual Analoge Scale (VAS) | Two years after DBS
  VAS measure of subjective or behavioral experience of back pain. Range 0-10 with higher scores indicating more severe symptoms.
  visual analog scale
Unified Parkinsons Disease Rating Scala (Part III Motor Examination) (UPDRS-Part III) | Two years after DBS
  The unified Parkinson's disease rating scale (UPDRS) to follow the longitudinal course of Parkinson's disease. Part III deals with motor experiences of daily living. It consists of 18 items. Each item has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe
Parkinsons Disease Questionaire 39 (PDQ-39) | Two years after DBS
  The PDQ-39 is a PD specific health status questionnaire comprising 39 items. Participants are requested to affirm one of five ordered response categories according to how often, due to their PD, they have experienced the problem defined by each item. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100 (100% more health problems).
Pelvic incidence (PI) | Two years after DBS
  The pelvic incidence (PI) corresponds to the angle between the perpendicular to the upper S1 level passing through its center and the line connecting this point to the axis of the femoral heads. Normal 45 ° to 65 °
Pelvit tilt (PT) | Two years after DBS
  The pelvic tilt (PT) is defined by the angle between the vertical and the line connecting the center of the sacral endplate to the axis of the femoral heads. Normal 3° to 18°
Sacral slope (SS) | Two years after DBS
  The sacral slope (SS) is defined by the angle between a line tangent to the upper S1 endplate and horizontal line. Normal -32° to -49°
Lumbar Lordisis (LL) | Two years after DBS
  Lumbar lordosis angle measures between the superior endplate of L1 and L5 inferior endplate. Norm 33.2 +/- 12.1 degrees
Mismatch of Pelvic incidence and LL (PI - LL) | Two years after DBS
  Difference between pelvic incidence and lumbar lordisis. Norm <10 degrees
Scoliosis | Two years after DBS
  Cobb Angle at a particular region of the vertebral column, when measured from the superior endplate of a superior vertebra to the inferior endplate of an inferior vertebra. No scoliosis <10°, mild scoliosis 10-30°, moderate scoliosis 30-45°, severe scoliosis >45°

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Spindler, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité University Medicine Department of Neurosurgery Campus Charité Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided